CLINICAL TRIAL: NCT02808052
Title: A Phase I, Open-Label, Single-Dose Trial To Determine The Safety And Pharmacokinetics Of Minocin (Minocycline) For Injection In Subjects With Renal Insufficiency
Brief Title: Evaluate Safety and Pharmacokinetics of Minocin (Minocycline) for Injection in Subjects With Renal Insufficiency
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision due to change in strategy
Sponsor: Rempex (a wholly owned subsidiary of Melinta Therapeutics, Inc.) (Industry)
Collaborators: Universitätsklinikum Köln (Other); Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Organization: Melinta Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDCO-MIN-16-03; 702 (Other: (IMI WP8B ID #))
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Renal Insufficiency, Acute; Renal Insufficiency, Chronic; Healthy Subjects
Keywords: Bacterial infections
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic; Bacterial Infections | interventions — Minocycline; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Minocin (minocycline) for Injection (Experimental): Minocin (minocycline) for Injection will be supplied as a sterile lyophilized powder in single-use 10-mL glass vials. Each vial contains 108 mg of minocycline hydrochloride equivalent to 100 mg of minocycline. Each cohort receives a single 200-mg dose of Minocin (minocycline) for Injection except for the hemodialysis therapy/end stage renal disease cohort, which receives two 200-mg doses.
  Interventions: Drug: Minocin (minocycline) for Injection

INTERVENTIONS:
Drug: Minocin (minocycline) for Injection — 200mg IV Minocin given over 1 hour
  Other Names: Minocin; minocycline

SUMMARY:
This is a Phase 1, open-label, single-dose study of the safety, tolerability, and pharmacokinetics of Minocin® (minocycline) for injection in subjects with renal insufficiency.

DETAILED DESCRIPTION:
The purpose of this study is to collect safety, tolerability, and pharmacokinetics (PK) data on a single dose of Minocin® (minocycline) for Injection in subjects with renal insufficiency and in subjects receiving hemodialysis therapy. The safety, tolerability, and PK data will support the compound as a potential clinical candidate in Europe and will inform the development of future Phase 2/3 studies.

ELIGIBILITY:
Inclusion Criteria:

1. A signed informed consent form, the ability to understand the study conduct and tasks that are required for study participation, and a willingness to cooperate with all tasks, tests, and examinations as required by the protocol, whether in the hospital or after discharge, for the duration of the study;
2. Healthy adult male or female between 18 and 85 years of age (inclusive) at the time of screening;
3. Subject has a body mass index (BMI) ≥ 18.5 kg/m2 and ≤ 45 kg/m2;
4. Pulse measured at screening/baseline must be within the ranges ≥ 45 to ≤ 115 beats per minute (bpm, taken after resting in a semi-recumbent position for at least 5 minutes);
5. Have sufficient peripheral vascular access, based on the Investigator's assessment, for all blood sample collections to take place;
6. Female subject is surgically sterile, postmenopausal, or if of childbearing potential, agrees to abstinence or to use at least 2 acceptable methods of birth control (e.g., prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, barrier methods, etc.) or male partner sterilization alone, between randomization and for 7 days after the completion of the study;

   Subjects with Renal Insufficiency:
7. Assessment of renal insufficiency for assignment to study groups will be based on measurements of estimated glomerular filtration rate calculated by the Modification of Diet in Renal Disease equation at the screening visit to determine eligibility;

   Subjects with Normal Renal Function:
8. Normal volunteers first matched by age (± 10 years), BMI (± 20%), and gender to the mean values of the moderate renal insufficiency group. Once the mild, moderate, and severe renal insufficiency groups are fully enrolled, the mean values of age, BMI, and gender will be calculated for the pooled renal insufficiency groups, and additional healthy subjects may be enrolled to match the pooled means;
9. Have a creatinine clearance (CrCl) ≥ 90 mL/min calculated using the Cockcroft Gault equation;

   Hemodialysis Subjects:
10. Receiving stable hemodialysis (Kt/V > 1.2) at least 3 times a week for at least 3 months, using an arteriovenous fistula or graft;
11. Otherwise considered to be clinically stable with respect to underlying renal impairment, as determined by the Investigator, and based upon a medical evaluation that includes a medical history, physical examination, laboratory tests, and electrocardiogram (ECG);
12. Have clinical laboratory test results that are considered clinically stable in the opinion of the Investigator, especially if the clinical abnormality or laboratory parameter is deemed associated with the subject's underlying renal impairment;
13. A stable medication regimen is required, defined as not starting new drug(s) or significant changes in dosage(s) within 14 days prior to administration of study drug, or during the conduct of the study. Changes of medications in hemodialysis subjects are subject to dialysis site protocols such that erythropoiesis-stimulating agents, iron, and vitamin D can be changed based on the then current subject status and dialysis unit standard practice and subject safety prior to screening.

Exclusion Criteria:

1. Has any condition, including findings in the medical history or in pre-study assessments, that are capable of altering the distribution, metabolism, or elimination of drugs or that constitute a risk or a contraindication for the participation in the study or completing the study; Subjects in the renal insufficiency groups will have consideration for the degree of renal insufficiency and presence of comorbidities;
2. Current evidence or history of malignancy, excluding basal cell carcinoma, in the 2 years prior to Day -1 (day before dosing) with no evidence of recurrence;
3. Blood or plasma donation within past 2 months;
4. Vigorous exercise from 48 hours prior to Day -1 until the day of discharge from the study;
5. Surgery within 48 hours prior to randomization or surgery planned during the study period;
6. Liver function abnormalities at screening (or Day -1) (defined by an elevation in bilirubin, aspartate aminotransferase, or alanine aminotransferase that is 1.5 x upper limit of normal of the normal range for subjects based on age and sex);
7. Females who are pregnant or nursing or who have a positive pregnancy test result;
8. Males who are unwilling to practice abstinence or use an acceptable method of birth control during the entire study period (i.e., condom with spermicide, where locally available);
9. Presence of known raised intracranial pressure;
10. Use of isotretinoin;
11. History of significant hypersensitivity or allergic reaction to tetracycline antibiotics;
12. History of seizures (e.g., epilepsy), head injury, or meningitis requiring ongoing anti-seizure medications;
13. Receipt of any investigational medication or investigational device during the last 30 days prior to randomization;
14. A corrected QT (Fridericia) > 500 msec or history of prolonged QT syndrome;
15. Use of products containing alcohol, caffeine, xanthine, or ephedrine within 48 hours before dosing;
16. Unable or unwilling, in the judgment of the Investigator, to comply with the protocol;
17. Subjects that have known active hepatitis B or C, or human immunodeficiency virus (HIV) infection or have known immune deficiency disease at screening;
18. Concurrent use of medications known to affect the elimination of serum creatinine (e.g., trimethoprim/sulfamethoxazole [Bactrim®] or cimetidine [Tagamet®]) and competitors of renal tubular secretion (e.g., probenecid) within 30 days prior to the first dose of study drug or anticipated need for these therapies through the last PK sample;
19. An employee of the Investigator or study center or sponsor, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center or the Sponsor, or a family member of the employee or the Investigator.

    Subjects with Renal Insufficiency:
20. Have a sitting systolic blood pressure (BP) > 180 mm Hg or < 90 mm Hg or have a sitting diastolic BP > 110 mm Hg or < 50 mm Hg at the screening visit;
21. Use of any other prescription or nonprescription drugs, vitamins, grapefruit/grapefruit juice, or dietary or herbal supplements within 14 days prior to Day -1 other than those listed below:

    1. Medications required to treat underlying renal disease or medical conditions related to renal disease are permitted;
    2. Oral contraceptives are permitted for birth control;
    3. Doses of concomitant medications (except hormonal contraceptives, hormone replacement therapy for females, and insulin) must be stable for 3 weeks prior to dosing on Day 1. Minor dose changes consistent with treatment practices may be permitted at the discretion of the Sponsor's Medical Monitor;
    4. Acetaminophen (≤ 1 g/day) and low dose acetylsalicylic acid (ASA, e.g., ≤ 325 mg per day) are permitted.

    Subjects with Normal Renal Function:
22. Abnormal and clinically significant findings on physical examination, medical history, serum chemistry, hematology, or urinalysis per Investigator discretion;
23. Have a sitting systolic BP > 150 mm Hg or < 90 mm Hg or have a sitting diastolic BP > 90 mm Hg or < 50 mm Hg at the screening visit;
24. CrCl < 90 mL/min calculated using the Cockcroft Gault equation;
25. Use of any prescription or nonprescription drugs, vitamins, grapefruit/grapefruit juice, or dietary or herbal supplements within 14 days prior to Day -1 other than those listed below:

    1. Oral contraceptives are permitted for birth control;
    2. Acetaminophen (≤ 1 g/day) and low dose ASA (i.e., ≤ 325 mg per day) are permitted.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Cornely, MD, Study Director — Universitätsklinikum Köln; Volker Burst, MD, PD, Principal Investigator — Universitätsklinikum Köln
Locations (1):
- University Hospital Cologne-Clinical Trial Center, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9 subjects were assigned to one of three groups (Mild, Moderate, or Severe) based on degree of renal impairment. All 9 subjects were enrolled in the study from 29-May-2017 to 17-Dec- 2017, at the Univ Hosp Cologne, Germany.
Pre-assignment Details: Following the change of ownership of Minocin IV from The Medicines Company to Melinta Therapeutics, the business decision was made to terminate this study prior to completion as Melinta.
Groups:
- Mild Renal Insufficiency: Mild renal insufficiency (eGFR 60-89 mL/min/1.73m2)
- Moderate Renal Insufficiency: Moderate renal insufficiency (eGFR 30 to < 60 mL/min/1.73m2)
- Severe Renal Insufficiency: Severe renal insufficiency (eGFR < 30 mL/min/1.73m2), not receiving hemodialysis (HD) therapy
Period: Overall Study
Arm/Group | Mild Renal Insufficiency | Moderate Renal Insufficiency | Severe Renal Insufficiency
Started | 4 | 3 | 2
Completed | 4 | 3 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Severe Renal Insufficiency: Severe renal insufficiency (eGFR < 30 mL/min/1.73m2), not receiving HD therapy
- Total: Total of all reporting groups
Arm/Group | Mild Renal Insufficiency | Moderate Renal Insufficiency | Severe Renal Insufficiency | Total
Number analyzed (Participants) | 4 | 3 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.25 (19.60) | 65.00 (11.53) | 54.00 (2.83) | 51.6 (17.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3
  Male | 2 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 3 | 2 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 4 | 3 | 2 | 9
Height [Mean (Standard Deviation); unit: cm] | 179.0 (4.08) | 176.67 (7.02) | 179.00 (1.41) | 178.22 (4.49)
Weight [Mean (Standard Deviation); unit: kg] | 80.98 (28.44) | 99.40 (2.08) | 111.05 (48.01) | 93.80 (27.59)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Intravenous Dose(s) of Minocin (Minocycline) for Injection Assessed by Number of Subjects With Adverse Events
Description: Safety and Tolerability: Subjects with mild, moderate, or severe renal insufficiency with any adverse events, any serious adverse events, any study related adverse events, and any adverse events with a fatal outcome.
Time Frame: Approximately 24 weeks
Population: All subjects (9) subjects who received at least one dose of study drug were included in the safety population used for safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Renal Insufficiency | Moderate Renal Insufficiency | Severe Renal Insufficiency
Number analyzed (Participants) | 4 | 3 | 2
Participants
  Number of subjects with any AE | 1 | 2 | 1
  Number of subjects with any SAE | 0 | 0 | 0
  Number of subjects with study related AE | 0 | 1 | 1
  Number subjects with AE leading to fatal outcome | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring from the time when first dose was administered up to the last follow-up visit (Day 6) where collected.
Arm/Group | Mild Renal Insufficiency | Moderate Renal Insufficiency | Severe Renal Insufficiency
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/4 | 2/3 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mild Renal Insufficiency (N=4) | Moderate Renal Insufficiency (N=3) | Severe Renal Insufficiency (N=2)
Headache (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Sputum Abnormal (Investigations) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Nightmare (Psychiatric disorders) | 0 | 1 | 0
Piloerection (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Early Termination of the study lead to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT02808052/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT02808052/SAP_001.pdf